CLINICAL TRIAL: NCT01111279
Title: Clinical Safety and Tolerability of gpASIT+TM Administered Subcutaneously in Absence or in Presence of DnaK Immunoregulating Adjuvant for the Prophylaxis of Seasonal Grass Pollen Rhinoconjunctivitis
Brief Title: Clinical Safety and Tolerability Study of gpASIT+TM and gpASIT+TM/Immunoregulating Adjuvant to Treat Seasonal Grass Pollen Rhinoconjunctivitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioTech Tools S.A. (Industry)
Responsible Party: Thierry Legon / CEO, BioTech Tools
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTT-gpASIT004
Record Dates: First submitted 2010-04-20; First posted 2010-04-27 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Seasonal Allergic Rhinoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo solution
- gpASIT+TM (Experimental)
  Interventions: Biological: gpASIT+TM
- gpASIT+TM/adjuvant (Experimental)
  Interventions: Biological: gpAST+TM/adjuvant

INTERVENTIONS:
Biological: gpASIT+TM — 1 subcutaneous injection every 7 days, during 29 days.
  Arms: gpASIT+TM
Biological: gpAST+TM/adjuvant — 1 subcutaneous injection every 7 days, during 29 days
  Arms: gpASIT+TM/adjuvant
Biological: Placebo solution — 1 subcutaneous injection every 7 days, during 29 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of gpASIT+TM administered subcutaneously in absence or in presence of an immunoregulating adjuvant in grass pollen allergic patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given written informed consent
* Age between 18 and 50 years
* The subjects are in good physical and mental health according to his/her medical history, vital signs, and clinical status
* Male or non pregnant, non-lactating female
* Females unable to bear children must have documentation of such in the CRF (i.e. tubule ligation, hysterectomy, or post menopausal (defined as a minimum of one year since the last menstrual period))
* Allergy diagnosis:

  * A history of seasonal allergic rhinoconjunctivitis (SAR) during the grass pollen season during at least during the two previous years
  * A positive skin prick test (wheal diameter ≥ 3 mm) to grass-pollen mixture
  * Specific IgE against grass pollen (RAST class 2 or IgE > 0.7 kU/l)
  * Asymptomatic to perennial inhalant allergens even if shown to be hypersensitive in a skin prick test.

Exclusion Criteria:

* Subjects with current or past immunotherapy (any time in the past)
* A history of hypersensitivity to the excipients
* Subjects requiring control medication against asthma (bronchodilator nebulised drugs or local or systemic corticosteroids)
* Subjects with documented evidence of acute or significant chronic sinusitis (as determined by investigator)
* Subjects with a history of hepatic or renal disease
* Subjects symptomatic to perennial inhalant allergens
* Subjects with rhinitis medicamentosa, non-specific rhinitis (to food dye, preservative agent…)
* Subject with malignant disease, autoimmune disease (and family medical history of autoimmune disease)
* Any chronic disease, which may impair the subject's ability to participate in the trial (i.e. severe congestive heart failure, active gastric or duodenal ulcer, uncontrolled diabetes mellitus, etc…)
* Subjects requiring beta-blockers medication
* Chronic use of concomitant medications that would affect assessment of the effectiveness of the trial medication (e.g. tricyclic antidepressants)
* Subject with febrile illness (> 37.5°C, oral)
* A known positive serology for HIV-1/2, HBs antigen or anti-HCV antibodies
* The subject is immunocompromised by medication or illness, has received a vaccine, corticoids or immunosuppressive medications within 1 month before trial entry
* Receipt of blood or a blood derivative in the past 6 months preceding trial entry
* Regular consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 4 weeks preceding the trial
* Any consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 1 week preceding the trial
* Use of long-acting antihistamines
* Female subjects who are pregnant, lactating, or of child-bearing potential and not protected from pregnancy by a sufficiently reliable method (OCs, IUD)
* Any condition which could be incompatible with protocol understanding and compliance
* Subjects who have forfeited their freedom by administrative or legal award or who are under guardianship
* Unreliable subjects including non-compliant subjects, subjects with known alcoholism or drug abuse or with a history of a serious psychiatric disorder as well as subjects unwilling to give informed consent or to abide by the requirements of the protocol
* Subjects without means of contacting the investigator rapidly in case of emergency, or not able to be contacted rapidly by the investigator
* Participation in another clinical trial and/or treatment with an experimental drug within 1 month of trial start
* Subjects who participated to trial BTT-gpASIT003 and were in the treated groups

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Clinical tolerability and safety of the treatment | 3 times during the treatment phase, at week 24 (the end of the study)
  The following parameters will be assessed : general physical status, vital signs, haematological parameters , general blood biochemistry parameters, all (serious) adverse, immunological analysis (total IgG, total IgE) and inflammatory parameters (CRP, sedimentation rate)

SECONDARY OUTCOMES:
Impact of gpASIT+TM on the immunological status of the subjects | visit 1, week 7, week 18 and week 24
  The following parameters will be assessed :
  * allergen-specific IgE, IgG, IgG4, IgA antibody concentrations,
  * adjuvant-specific IgG antibody concentrations,
  * lymphoproliferation and production of IL-10 in allergen and adjuvant stimulated PBMC.
Impact of gpASIT+TM on the clinical status of the subjects | 1 May - 15 August 2010
  The following parameters will be assessed (during the pollen season following treatment):
  * daily average allergic symptom score,
  * daily average allergic medication score,
  * number of "well-days",
  * Visual Analogue Scale .

CONTACTS AND LOCATIONS:
Overall Officials: Jan Ceuppens, Professor, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Gasthuisberg, Leuven, Belgium